CLINICAL TRIAL: NCT02659215
Title: A Prospective, Randomized, Active Treatment-controlled, Evaluator-blinded Multicenter Study to Establish the Superiority of Hyalofast® With BMAC in the Treatment of Articular Knee Cartilage Defect Lesions in Comparison to Control
Brief Title: HyaloFAST Trial for Repair of Articular Cartilage in the Knee
Acronym: FastTRACK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hyalofast 15-01
Record Dates: First submitted 2016-01-14; First posted 2016-01-20 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Defect of Articular Cartilage
Keywords: Hyaluronic Acid; Cartilage Repair; Knee
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyalofast with BMAC (Experimental): A hyaluronan-based scaffold (Hyalofast®) is utilized together with autologous bone marrow aspirate concentrate (BMAC) in a one-step arthroscopic/mini-arthrotomic procedure.
  Interventions: Device: Hyalofast
- Microfracture (Active Comparator): Microfracture is an arthroscopic surgical technique involving placement of microfracture penetrations within the cartilage defect to provide stem cells and growth factors from the bone marrow to aid cartilage repair.
  Interventions: Procedure: Microfracture

INTERVENTIONS:
Device: Hyalofast — Implantation of Hyalofast scaffold with autologous bone marrow aspirate concentrate via arthroscopy/mini-arthrotomy.
  Arms: Hyalofast with BMAC
Procedure: Microfracture — Microfracture is a well-established arthroscopic surgical technique for cartilage repair which involves several systematic steps, including debridement to a stable cartilage margin, careful removal of the calcified cartilage layer, and homogeneous placement of microfracture penetrations within the cartilage defect, with resultant complete defect fill by a well-anchored clot
  Arms: Microfracture

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Hyalofast® scaffold with bone marrow aspirate concentrate (BMAC) compared to microfracture in the treatment of symptomatic cartilage defects of the knee.

DETAILED DESCRIPTION:
* Prospective, randomized, active treatment-controlled, evaluator-blinded (radiologist reviewer and physician evaluator) multicenter study (up to 40 sites in the US and EU).
* All subjects that meet preoperative screening eligibility criteria will be randomized to treatment with Hyalofast® with BMAC or Microfracture.
* Hyalofast® is a sterile, biodegradable non-woven pad (2 x 2 cm or 5 x 5 cm) that is composed of HYAFF-11®, a benzyl ester of hyaluronic acid. Hyalofast® acts as a biodegradable support for the autologous bone marrow aspirate concentrate. Hyalofast® is soft and conformable and can easily be cut to fit the lesion size.
* Autologous bone marrow is harvested from the subject intraoperatively during the Index Procedure. Approximately 60 mL of bone marrow will be aspirated from the subject's iliac crest using the SmartPrep 2 Bone Marrow Processing Pack. The cellular rich portion will be concentrated via the SmartPrep BMAC 2 Centrifuge System at point-of-care to provide 7 mL of bone marrow aspirate concentrate (BMAC). 1 - 2 mLs will be used for post-procedure testing of total nucleated cells, cell viability, and sterility.
* Hyalofast® with BMAC is implanted during either a standard knee arthroscopy or min-arthrotomy depending upon surgeon preferences and intra-operative findings. The lesion to be treated will be debrided to a stable cartilage margin. The defect will be sized and Hyalofast® will be cut to fit the lesion area. If necessary, more than one Hyalofast® pad can be overlapped to cover the lesion. 2 mL of BMAC will be loaded per Hyalofast® scaffold and then implanted to cover the defect. Hyalofast® with BMAC readily adheres to the site of application, but, if necessary, can be secured to the defect margins with an FDA-approved fibrin glue.
* All subjects will be assessed at intervals post-procedure (1 month, 3 months, 6 months, 12 months, 24 months, and 36 months).
* Subjects will be required to follow a strict pre-specified post-surgery rehabilitation protocol specific to the defect location.
* Measures to assess effectiveness will be conducted at follow-ups, with the primary effectiveness endpoint assessment done at the 24 month timepoint.
* Evaluators doing efficacy assessments of the subject and administering subject-reported outcome instruments will be blinded to the treatment.
* Safety will be assessed by the collection of adverse events at all timepoints.
* Magnetic Resonance Imaging (MRI) will be conducted at Screening, 1 month, 12 months, 24 months, and 36 months. Evaluation of the MRIs, including the MOCART score, will be done by blinded radiologist reviewers. The one month MRI will be used as the baseline MRI for evaluation of treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female, between 18 and 60 years of age
2. Patient's body mass index (BMI) is <35 kg/m2
3. Patient has a symptomatic lesion of the femoral condyle (medial and/or lateral) or femoral trochlea that is between 1.5 - 6 cm2 on screening images confirmed by the independent radiologist
4. The symptomatic lesion is classified as International Cartilage Repair Society (ICRS) grade 3 or 4
5. Patient agrees to actively participate in a strict rehabilitation protocol and follow-up program
6. Patient is using only nonsteroidal anti-inflammatory drugs or acetaminophen/paracetamol during the month before signing the informed consent form to treat knee pain
7. Patient is willing and able to provide informed consent and comply with study requirements
8. Patient, if woman of childbearing potential, must have a negative pregnancy test at Screening, cannot be lactating and is willing to use adequate contraception for the first 12 months of the study after the last surgery
9. Patient has ability to consistently rate knee pain and function as demonstrated by completion of total KOOS score
10. Patient has a minimum of 45 out of 100 Visual Analogue Scale (VAS) score for index knee pain when remembering index knee pain when not on medication and when active
11. Patient is willing to use other pain medication rather than Non-steroidal Anti-inflammatory Drugs (NSAIDS) for 6 months post-surgery (e.g. acetaminophen, or narcotic analgesics, if prescribed). Post-surgical use of aspirin for clot prevention is acceptable.
12. Patient is willing to restrict pain medication after 6 months post-surgery to NSAIDs or acetaminophen/paracetamol only through the end of the trial
13. Patient must have Hematocrit ≥ 28.0%; White Blood Cell count ≤ 14,000; Platelet Count ≥ 50,000; Creatinine ≤ 2.0 mg/dL; and International Normalized Ratio (INR) ≤ 1.6

Exclusion Criteria:

1. Major concomitant cartilage lesions which require extensive surgical treatment. (Lesions such as minor loose bodies, small debris fragments, small cartilage fragments or prominent knee fat pad are allowed. These lesions may be treated with debridement).
2. Presence of a kissing bipolar lesion that is apposed to the index lesion and is deeper than Grade 2 (ICRS classification) as determined by MRI. (Presence of a kissing (bipolar) lesion that is apposed to the index lesion and is deeper than Grade 2 and is discovered under arthroscopy are allowed). The non-index lesion, if indicated for treatment, should be treated with the study assigned treatment of the index lesion.
3. Diagnosed advanced osteoarthritis as demonstrated by a Kellgren-Lawrence grade of 3 or 4 in the index knee
4. Complex ligamentous instability of the index or contralateral knee. (Previous reconstructions of Anterior Cruciate Ligament (ACL) or Posterior Cruciate Ligament (PCL) are allowed, of either the index or contralateral knee, if instability is not present. Grade 1 ligamentous injury are allowed)
5. Infections or skin diseases at target knee joint
6. Osteochondritis dissecans (OCD)
7. Patients requiring meniscal arrow or meniscal sutures
8. Previous meniscal transplant in the index knee
9. Patients with previous total or functional meniscectomy. (Patients with a previous partial meniscectomy and a meniscus that is considered biomechanically functional are allowed)
10. Varus or valgus malalignment exceeding 10° in either knee
11. Patient requiring concomitant surgical procedures at the time of Index Procedure such as osteotomies (e.g. high tibial valgus and/or patellar realignment osteotomy), bone subchondral perforation, ligament surgery, meniscal surgeries etc.
12. Previous cartilage repair procedure (microfracture, Osteochondral autograft transplantation system (OATS) or Autologous Chondrocyte Implantation (ACI) with or without use of a scaffold (matrix) in the index knee
13. Previous failed microfracture procedure in index knee. (Previous history of microfracture in the contralateral knee is allowed)
14. Known hypersensitivity (allergy) to hyaluronate
15. Contraindication(s) to microfracture surgery
16. Hyaluronic acid intra-articular injections into the index knee within the last 90 days before signing informed consent
17. Corticosteroid therapy by systemic or intra-articular route within the last 60 days before informed consent or intramuscular or oral corticosteroids within the last 30 days before informed consent.
18. Uncontrolled diabetes
19. Any concomitant painful or disabling disease of the spine, hips, or lower limbs, including the contralateral knee, that would interfere with evaluation of the index knee
20. Any clinically significant or symptomatic vascular or neurologic disorder of the lower extremities
21. Any evidence of the following diseases in the index knee: septic arthritis; inflammatory joint disease; gout; recurrent episodes of pseudogout; Paget disease of bone; ochronosis; acromegaly; hemochromatosis; Wilson disease; primary osteochondromatosis; heritable disorders; collagen gene mutations
22. Rheumatoid arthritis or gouty arthritis
23. Current diagnosis of osteomyelitis
24. Any result from screening blood work (including complete blood count, Prothrombin Time (PT)/Partial Thromboplastin Time (PTT)/INR, liver function, and creatinine) that exceeds 1.5x the upper limit of normal or is below 0.5x the lower limit of normal.
25. Diagnosed musculoskeletal cancer or any diagnosed cancer, other than musculoskeletal if not on long term remission (e.g. at least 5 years or negative biopsy at last exam), except basal cell carcinoma
26. Alcohol and drug (including medication) abuse
27. Patients who are at higher risk for post-surgical bleeding (e.g., bleeding disorder; taking anticoagulants except low dose aspirin) or post-surgical infection (e.g., taking immunosuppressants; have a severe infection or a history of serious infection)
28. Contraindications to MR imaging
29. Patient is currently receiving workman's compensation or disability or is in litigation for workman's compensation or disability claims
30. Participation in concurrent trials or in previous trial within 90 days of signing informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Superiority of Hyalofast with Bone Marrow Aspirate Concentrate (BMAC) vs. Microfracture for % Change in Knee injury and Osteoarthritis Outcome Score (KOOS) Pain Score | 2 years post-surgery
  Co-primary endpoint
Superiority of Hyalofast with Bone Marrow Aspirate Concentrate (BMAC) vs. Microfracture for % Change in International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Score | 2 years post-surgery
  Co-Primary Endpoint

SECONDARY OUTCOMES:
Superiority of Hyalofast® with autologous BMAC vs. Microfracture for change in MRI MOCART Score from baseline to two years post-surgery | 2 years post-surgery
Superiority of Hyalofast® with autologous BMAC vs. Microfracture for change in Evaluator Global Assessment from baseline to two years post-surgery | 2 years post-surgery
Superiority of Hyalofast® with autologous BMAC vs. Microfracture in change in individual KOOS subscales from baseline to two years post-surgery | 2 years post-surgery
Superiority of Hyalofast® with autologous BMAC vs. Microfracture in change in IKDC Knee Examination Form domains from baseline to two years post-surgery | 2 years post-surgery
The incidence, timing, severity, and relationship to treatment of all Adverse Events (AE), will be collected for all participants. | 3 years post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Gobbi, MD, Principal Investigator — OASI Bioresearch Foundation
Locations (48):
- United States (18):
  - Physicians Research Group, Tempe, Arizona
  - Axis Clinical Trials, Los Angeles, California
  - Kerlan-Jobe Orthopedic Clinic, Los Angeles, California
  - BioSolutions Clinical Research Center, San Diego, California
  - New Hope Research Development, Tarzana, California
  - Orthopedic Foundation, Stamford, Connecticut
  - Paramount Trials, LLC, Miami, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - OrthoIllinois, Rockford, Illinois
  - Bone and Joint Clinic of Baton Rouge, Baton Rouge, Louisiana
  - Covington Orthopedic and Sports Medicine Institute, Covington, Louisiana
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - New York Presbyterian Hospital, New York, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Penn Medicine, Philadelphia, Pennsylvania
  - Austin Ortho Biologics / Seton Medical Center Austin, Austin, Texas
  - Baylor Scott & White, Temple, Texas
  - Epic Medical Research, Murray, Utah
- Austria (8):
  - University Hospital Tulln, Tulln, Lower Austria
  - Kepler University Clinic, Linz, Upper Austria
  - Krankenhaus der Barmherzigen Schwestern, Ried, Upper Austria
  - Medical University of Graz, Graz
  - Universtitatsklinkik Krems, Krems
  - Medical University of Vienna, Vienna
  - Evangelisches Krankenhaus, Vienna
  - Private Hospital Doebling, Vienna
- Estonia (2):
  - Ortopeedia Arstid AS, Tallinn
  - North Estonia Medical Center, Tallinn
- Hungary (9):
  - Health Center of Downtown-Lipotvaros, Orthopedic Outpatient Clinic (Belvárosi-Lipótvárosi Egészségügyi Szolgálat Ortopeadia), Budapest
  - Semmelweis Egyetem Orthopaedic Clinic (Ortopédiai Klinika), Budapest
  - Uzsoki Hospital, Department of Traumatology, Budapest
  - Jutrix Medical Llc, Budapest
  - Menta Egeszsegkozpont Kft., Budapest
  - Magyar Honvedseg, Egeszseugyi Kozpont, Balesteti Sebeszeti Osztaly, Budapest
  - DE KK Ortopediai Klinika, Debrecen
  - Somogy Megyei Kaposi Mór Oktatókórház, Kaposvár
  - Kastelypark Klinka, Tata
- Indonesia (2):
  - Medistra Hospital, Jakarta
  - Royal Progess Hospital, Jakarta
- Italy (3):
  - Instituto Ortopedico Rizzoli, Bologna
  - A.O. Universitaria San Martino Monoblocco, Genova
  - University Federico II, Naples
- Lithuania (2):
  - AB "Ortopedijos technika", Kaunas
  - Vilnius University Hospital Santaros klinikos, Vilnius
- Mexico (3):
  - Desarrollo Ético en Investigación Clínica S.C., Guadalajara
  - Cruz Roja Mexicana (Hospital de Ortopedia de la Cruz Roja Mexicana), Mérida
  - Hospital Universitario Dr. José Eleuterio González, Monterrey
- De La Salle Medical and Health Sciences Institute, Cavite, Philippines

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah SS, Lee S, Mithoefer K. Next-Generation Marrow Stimulation Technology for Cartilage Repair: Basic Science to Clinical Application. JBJS Rev. 2021 Jan 19;9(1):e20.00090. doi: 10.2106/JBJS.RVW.20.00090. PMID 33512974